CLINICAL TRIAL: NCT00003132
Title: Phase I Study of Bryostatin-1 (NSC 339555) and Cisplatin in Advanced Malignancies
Brief Title: Bryostatin 1 Plus Cisplatin in Treating Patients With Metastatic or Unresectable Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000065897; NYU-9709; NCI-T97-0058
Record Dates: First submitted 1999-11-01; First posted 2004-04-07 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2009-11

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — bryostatin 1; Cisplatin

INTERVENTIONS:
Drug: bryostatin 1
Drug: cisplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of bryostatin 1 plus cisplatin in treating patients who have metastatic or unresectable cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and dose limiting toxicity of bryostatin 1 in combination with cisplatin in patients with advanced malignancy. II. Determine the recommended phase II doses of bryostatin 1 and cisplatin in both a 21 day and 14 day course, based on toxicity, effect on protein kinase C activity, and pharmacokinetics, in this patient population. III. Determine the pharmacokinetics of bryostatin 1 in these patients. IV. Identify any objective tumor responses arising from treatment in these patients.

OUTLINE: This is a dose escalation study of bryostatin 1. Cohorts 1-7: Patients receive cisplatin IV over 1 hour on day 1 of the first course. Subsequent courses repeat every 21 days with bryostatin 1 IV over 24 hours on day 1 and cisplatin IV over 1 hour on day 2 in the absence of disease progression or unacceptable toxicity. Cohorts 8-10: Patients receive cisplatin as in cohorts 1-7. Subsequent courses repeat every 21 days with bryostatin 1 IV over 1 hour followed by cisplatin on day 1. Cohort 11: Patients receive bryostatin 1 and cisplatin as in cohorts 8-10. Cohorts of 3-6 patients receive escalating doses of bryostatin 1 or cisplatin until the maximum tolerated dose (MTD) of is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience DLT. The recommended phase II dose (RPTD) is defined as the dose preceding the MTD. After the RPTD is determined for the 21 day schedule, cohorts of patients receive escalating doses of bryostatin and constant doses of cisplatin on a 14 day schedule. The MTD14 and RPTD14 are determined in the same manner as above. Patients are followed for 6 months.

PROJECTED ACCRUAL: A total of 36-72 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic or unresectable malignant disease Prior brain metastases with no residual signs or symptoms or medications allowed

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) AST/ALT no greater than 2.5 times ULN Alkaline phosphatase no greater than 2.5 times ULN Renal: Creatinine no greater than 1.5 mg/dL Other: Not pregnant or nursing Fertile patients must use effective contraception No concurrent condition that would preclude study No psychological, familial, sociological, or geographical condition that might compromise medical follow up No neuropathy greater than grade 1, including hearing loss

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 3 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas)and recovered Prior cisplatin allowed Endocrine therapy: Not specified Radiotherapy: At least 2 weeks since prior radiotherapy Prior radiotherapy for brain metastases allowed Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-01; Primary Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco M. Muggia, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Pavlick AC, Wu J, Roberts J, Rosenthal MA, Hamilton A, Wadler S, Farrell K, Carr M, Fry D, Murgo AJ, Oratz R, Hochster H, Liebes L, Muggia F. Phase I study of bryostatin 1, a protein kinase C modulator, preceding cisplatin in patients with refractory non-hematologic tumors. Cancer Chemother Pharmacol. 2009 Sep;64(4):803-10. doi: 10.1007/s00280-009-0931-y. Epub 2009 Feb 17. PMID 19221754
- [Result] Pavlick AC, Hamilton A, Liebes L, et al.: Bryostatin 1 and cisplatin: a phase I and pharmacodynamic study. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-328, 2001.